CLINICAL TRIAL: NCT02540785
Title: Comparison of Early Changes in Ocular Surface and Inflammatory Mediators Between Lenticule Extraction and Small-Incision Lenticule Extraction
Brief Title: Early Changes Between Lenticule Extraction and Small-Incision Lenticule Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xingwu Zhong, MD PhD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-005
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Myopia; Astigmatism
Keywords: Refractive Surgical Procedures; small-incision lenticule extraction; lenticule extraction; inflammatory mediators
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Tobramycin; Dexamethasone; Tobramycin, Dexamethasone Drug Combination; methylacetylene; Levofloxacin; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lenticule extraction (Experimental): The patients in this group chose to receive the lenticule extraction surgery.
  Interventions: Procedure: lenticule extraction
- small-incision lenticule extraction (Experimental): The patients in this group chose to receive the small-incision lenticule extraction surgery.
  Interventions: Procedure: small-incision lenticule extraction

INTERVENTIONS:
Procedure: lenticule extraction — Four femtosecond incisions were created in succession: the posterior surface of the refractive lenticule (spiral in), the lenticule border, the anterior surface of the refractive lenticule (spiral out), and the corneal flap in the superior region. After the suction was released, the flap was opened using a thin, blunt spatula and the free refractive lenticule was subsequently grasped with a forceps and extracted, after which the flap was repositioned carefully
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon); 0.5% levofloxacin (Cravit, Santen); sodium hyaluronate (HYCOSAN,URSAPHARM Arzneimittel GmbH)
  Arms: lenticule extraction
Procedure: small-incision lenticule extraction — Four femtosecond incisions were created in succession: the posterior surface of the refractive lenticule (spiral in), the lenticule border, the anterior surface of the refractive lenticule (spiral out), make a small incision
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon); 0.5% levofloxacin (Cravit, Santen); sodium hyaluronate (HYCOSAN,URSAPHARM Arzneimittel GmbH)
  Arms: small-incision lenticule extraction

SUMMARY:
The aim is to evaluate the short-term changes in ocular surface measures and tear inflammatory mediators after lenticule extraction (FLEx) and small-incision lenticule extraction (SMILE) procedures.

DETAILED DESCRIPTION:
The use of femtosecond (FS) laser has become one of the most significant technological advancements in refractive surgery. A breakthrough FS laser-assisted myopic and myopic astigmatic correction procedure can now be performed using a prototype femtosecond system. This first all-in-one FS-laser system was designed to perform the refractive lenticule extraction (ReLEx) procedures, femtosecond lenticule extraction (FLEx) and small-incision lenticule extraction (SMILE). In FLEx, a corneal flap is created by the FS laser (similar to LASIK) and lifted, allowing lenticule removal. For SMILE, a truly without flap procedure, only a small-2-4mm- incision is made, through which the lenticule is removed.

Ocular surface disruption during corneal refractive surgery is commonly considered to be closely related to the development of dry eye. Multiple etiologies contribute to this ocular surface disruption, including the flap creation and stromal ablation involved in previous refractive surgery techniques. Corneal nerve damage has been considered the main cause of dry eye, due to disrupted afferent sensory nerves, reduced blink reflex, and increased tear evaporation leading to tear film instability. In addition, postoperative inflammatory mediator fluctuations are also a key factor related to ocular surface damage. Extensive research has described the effects of cytokines, chemokines and growth factors in modulating corneal wound healing, cell migration, and apoptosis on the ocular surface after refractive surgery.

For both FLEx and SMILE, stromal ablation has been replaced by refractive lenticule removal. In terms of corneal flap formation, FLEx still requires an epithelial-stromal flap, while SMILE employs only a small incision to extract the lenticule. Hence, the investigators hypothesize that SMILE will have less effect on patients' ocular surface markers and inflammatory mediators, compared to FLEx. In support of this hypothesis, previous studies have reported that more damage to the sub-basal nerve plexus of the cornea and more changes in ocular surface evaluations were found after FLEx than after SMILE. In this study, the investigators have focused on postoperative changes to tear inflammatory mediators and the relationship of FLEx and SMILE to dry eye.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years(range from 18 year to 25 years); corneal thickness 500 μm with calculated residual stromal bed after treatment greater than 300 μm; preoperative spherical equivalent refraction between
* 2.00 diopter (D) and -6.50 D; preoperative cylindrical equivalent refraction between -0.25 D and -1.50 D; preoperative corneal curvature from 41.0 D to 46.0 D with a regular topographic pattern, verified with an Atlas topographer; monocular best corrected visual acuity of 20/20 or better and stable refractive error (less than 0.5 D change) for 24 months before surgery

Exclusion Criteria:

* systemic disease that contraindicated the surgery (such as diabetes, glaucoma and systemic collagen vascular disease); corneal abnormality or disease; a history of tear supplement usage or contact lens wear during the past year

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
scale of Schirmer I test | up to 1month after surgery
scale of corneal fluorescein staining | up to 1month after surgery
scale of noninvasive tear breakup time | up to 1month after surgery
questionnaire of ocular surface disease index | up to 1month after surgery
scale of central corneal sensitivity | up to 1month after surgery
scale of tear meniscus height | up to 1month after surgery
concentration of Interleukin-1α | up to 1month after surgery
concentration of tumor necrosis factor-α | up to 1month after surgery
concentration of nerve growth factor | up to 1month after surgery
concentration of interferon-γ | up to 1month after surgery
concentration of transforming growth factor-β1 | up to 1month after surgery
concentration of matrix metalloproteinase-9 | up to 1month after surgery

SECONDARY OUTCOMES:
Correlation Between Inflammatory Mediators and Ocular Surface Changes | up to 1month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xingwu Zhong, MD PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University

REFERENCES:
- [Derived] Zhang C, Ding H, He M, Liu L, Liu L, Li G, Niu B, Zhong X. Comparison of Early Changes in Ocular Surface and Inflammatory Mediators between Femtosecond Lenticule Extraction and Small-Incision Lenticule Extraction. PLoS One. 2016 Mar 3;11(3):e0149503. doi: 10.1371/journal.pone.0149503. eCollection 2016. PMID 26937680